CLINICAL TRIAL: NCT04882800
Title: Evaluation of Fitting Modification for Extended Wear Technology
Brief Title: Evaluation of Extended Wear Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SRF-72
Record Dates: First submitted 2021-05-04; First posted 2021-05-12 (Actual); Results first posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-07

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: Participants will be fit with commercially available extended wear hearing aid device A in the right ear and extended wear hearing aid with fitting modifications device B in the left ear for two weeks (first intervention); then fit with extended wear hearing aid with fitting modifications device B in the right ear and commercially available extended wear hearing aid device A in left ear for two weeks (second intervention). There will be no washout period.
Masking Description: Participants will not know which device is in each ear, only that they are being fit with Lyric devices.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- First Intervention (Experimental): Participants will be fit with currently available Lyric extended wear hearing aid device A in right ear and Lyric extended wear hearing aid with fitting modification device B in left ear for 14 days (Day 1 - Day 14 of study). They will then switch and be fit with Lyric extended wear hearing aid with fitting modification device B in the right ear and the commercially available Lyric device A in the left ear for 14 days (Day 15-Day 28 of study)
  Interventions: Device: Lyric extended wear hearing aid device A; Device: Lyric extended wear hearing aid with fitting modification device B

INTERVENTIONS:
Device: Lyric extended wear hearing aid device A — Current commercially available extended wear hearing aid
Device: Lyric extended wear hearing aid with fitting modification device B — Extended wear hearing aid with fitting modifications

SUMMARY:
Evaluating the efficacy and effectiveness of an advancement in the fitting characteristics of extended wear technology with the commercially available device as a comparator.

DETAILED DESCRIPTION:
A interventional study in which participants will be fit with the commercially available device in one ear and the experimental device in the opposite ear. After two weeks, the devices will be switched so that the participant has worn each device in each ear for a total of 2 weeks. Participants will be blinded as to which device they are wearing in each ear. Comfort and sound quality will be assessed for each device prior to removing from ears.

ELIGIBILITY:
Inclusion Criteria:

* Mild, Moderate and Moderate Severe Hearing loss
* Previous extended wear technology users who rejected or cancelled trials due to discomfort, feedback, migration, or poor sound quality due to fit issues

Exclusion Criteria:

* Participants who can only wear a size XXS (extra-extra small) extended wear device
* asymmetrical hearing loss
* other diagnosis that may cause hearing fluctuation
* inability to tolerate physical fit of Lyric devices
* inability to be seen for four lab visits

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Seitz-Paquette, AuD, Principal Investigator — Sonova AG
Locations (1):
- Main Line Audiology Consultants, Narberth, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Participants will be fit with commercially available Lyric extended wear hearing aid device A in right ear and Lyric extended wear hearing aid with fitting modification device B in left ear for two weeks (Day 1- Day 14 of study). They will then switch and be fit with device B in the right ear and device A in the left ear for two weeks (Day 15-Day 28 of study).
  Lyric extended wear hearing aid device A: Current commercially available extended wear hearing aid
  Lyric extended wear hearing aid with fitting modification device B: Extended wear hearing aid with fitting modifications
Period: Device A Right Ear/Device B Left Ear
Arm/Group | Intervention
Started | 15
Completed | 15
Not Completed | 0
Period: Device B Right Ear/Device A Left Ear
Arm/Group | Intervention
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Experienced hearing aid users
Groups:
- All Study Participants: All participants who were fit with hearing aid device A in right ear and hearing aid device B in left ear Day 1 to Day 14 of study, and then fit with device B in the right ear and device A in the left ear Day 15 to Day 28 of study.
  Lyric extended wear hearing aid device A: Current commercially available extended wear hearing aid
  Lyric extended wear hearing aid with fitting modification device B: Extended wear hearing aid with fitting modifications
Arm/Group | All Study Participants
Number analyzed (Participants) | 15
Age, Continuous [Mean (Full Range); unit: years] | 68 [34 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Subjective Questionnaire of Comfort
Description: Subjective ratings of comfort of each device in the ear, on a scale from 0 (very comfortable) to 10 (very uncomfortable/painful). No statistical analysis was planned for this measure.
Time Frame: Two weeks after fitting device A in right ear/device B in left ear (Day 14 of study), and two weeks after fitting device A in left ear/device B in right ear (Day 28 of study-final appointment)
Population: All participants who were fit with commercially available Lyric extended wear hearing aid device A in right ear and Lyric extended wear hearing aid device B in left ear Day 1- Day 14, and who were fit with extended wear hearing aid device B in right ear and commercially available hearing aid device A in left ear Day 15 to Day 28 of study.
Measure: Median (Full Range); unit: score on a scale
Units Other Than Participants: Ears
Groups:
- Intervention: Participants fit with commercially available Lyric extended wear hearing aid device A in right ear and Lyric extended wear hearing aid with fitting modification device B in left ear for two weeks,(Day 1 to Day 14 of study). They will then switch and be fit with device B in right ear and device A in left ear for two weeks (Day 15-Day 28 of study).
  Lyric extended wear hearing aid device A: Current commercially available extended wear hearing aid
  Lyric extended wear hearing aid with fitting modification device B: Extended wear hearing aid with fitting modifications
Arm/Group | Intervention
Number analyzed (Participants) | 15
Number analyzed (Ears) | 30
score on a scale
  Comfort Rating of Device A | 0 [0 to 7]
  Comfort Rating of Device B (investigational device) | 0 [0 to 10]

2. Primary Outcome: Subjective Ratings of Occlusion With Both Devices
Description: Subjective ratings on how plugged participants' ears felt with each device in ear,on scale from 0 (not at all) to 10 (extremely plugged/cannot tolerate)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Units Other Than Participants: Ears
Groups:
- Intervention: Participants fit with commercially available Lyric extended wear hearing aid device A in right ear and Lyric extended wear hearing aid with fitting modification device B in left ear for two weeks,(Day 1 to Day 14 of study). They will switch and wear device B in right ear and device A in left ear for two weeks (Day 15-Day 28 of study).
  Lyric extended wear hearing aid device A: Current commercially available extended wear hearing aid
  Lyric extended wear hearing aid with fitting modification device B: Extended wear hearing aid with fitting modifications
Arm/Group | Intervention
Number analyzed (Participants) | 15
Number analyzed (Ears) | 30
score on a scale
  Occlusion Rating with Device A | 0 [0 to 8]
  Occlusion Rating with Device B (fitting modification) | 0 [0 to 10]

ADVERSE EVENTS:
Time Frame: 4 weeks
Groups:
- First Intervention (Device A in Right Ear and Device B in Left Ear): Participants fit with commercially available Lyric extended wear hearing aid device A in right ear and Lyric extended wear hearing aid with fitting modification device B in left ear for two weeks,(Day 1 to Day 14 of study).
  Lyric extended wear hearing aid device A: Current commercially available extended wear hearing aid
  Lyric extended wear hearing aid with fitting modification device B: Extended wear hearing aid with fitting modifications
- Second Intervention (Device B in Right Ear and Device A in Left Ear): Participants fit with Lyric extended wear hearing aid with fitting modification device B in right ear and commercially available Lyric extended wear hearing aid device A in left ear for two weeks,(Day 15 to Day 28 of study).
  Lyric extended wear hearing aid device A: Current commercially available extended wear hearing aid
  Lyric extended wear hearing aid with fitting modification device B: Extended wear hearing aid with fitting modifications
Arm/Group | First Intervention (Device A in Right Ear and Device B in Left Ear) | Second Intervention (Device B in Right Ear and Device A in Left Ear)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-20): https://cdn.clinicaltrials.gov/large-docs/00/NCT04882800/Prot_SAP_000.pdf